CLINICAL TRIAL: NCT07151365
Title: Plant-based Diets and Healthy Aging - the Tzu Chi Aging Study (TCAS)
Brief Title: Plant-based Diets and Healthy Aging
Acronym: TCAS
Status: Enrolling by invitation | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Other Study IDs: EC1131206; IRB approval number (Other: NHRI Taiwan Institutional Review Board (IRB))
Record Dates: First submitted 2025-08-17; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy Aging; Sarcopenia; Frailty; Cognitive Decline
Keywords: Vegetarian diets; Plant-based diets; Healthy aging; Cognitive decline; Sarcopenia; Frailty
MeSH Terms: conditions — Sarcopenia; Frailty; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This prospective study investigates the health effects of vegetarian and plant-based diets in middle-aged and older adults in Taiwan, specifically, recruiting 5000 Tzu Chi volunteers. Previous Tzu Chi cohorts found vegetarian diets were protectively associated with incidences of diabetes, stroke, gout, cataracts, insomnia, and gallstones, while reducing healthcare costs. The study also aims to clarify dietary patterns-particularly plant-based and vegetarian diets-and determine how potential deficiencies or excesses of various nutrients influence common aging-related health issues, including healthy cognitive decline, sarcopenia, and the risk of age-related diseases, in order to inform dietary and lifestyle recommendations that promote healthy aging and maintain physical function.

DETAILED DESCRIPTION:
This study establishes a new cohort to investigate the role of vegetarian and plant-based diets in healthy aging, integrating functional, nutritional, and genetic data. The primary objective is to clarify how dietary patterns and nutrient intake influence aging-related health conditions, including sarcopenia, cognitive function, physical function, and psychological well-being, and investigate how the associations between diet and these health conditions may be modified by genetic risk factors.

Participants are Tzu Chi volunteers aged 40 years and older who undergo comprehensive health evaluations at Dalin Tzu Chi Hospital every three years. This population consists of a uniquely high proportion of vegetarians, non-smoking non-alcohol drinking individuals, and older adults who are active in communities and social engagement and community services; providing a unique opportunity to examine the role of plant-based diets and community services on aging related conditions without confounding by smoking and alcohol. Diet data are collected through a previously validated food frequency questionnaire, a short newly developed questionnaire - Taiwan Diet Quality Calculator - that will be validated within a subcohort of the current study, and food diaries for participants who are willing to provide such details. Nutritional biomarkers (e.g., serum vitamin B12, vitamin D, skin carotenoids), along with routine health examination values (complete blood counts, lipid profiles, renal and liver functions, bone mineral density) will also be collected. When funding permits, genome-wide genotyping, metabolomics, and other aging-related biomarkers will also be examined.

For cohort follow-up, study participants will be invited back for follow-up health examination every three years. In addition, data will also be linked to National Health Insurance Claim database, National Cancer registry, and National Mortality Registry in Taiwan to further ascertain relevant health outcomes.

By integrating comprehensive dietary assessments, nutritional biomarkers, health examination and genetic data, and aging-related functional outcomes, this cohort will provide an unique opportunity to examine dietary patterns, nutrient requirements, and lifestyle that best support healthy aging. The inclusion of genomic and metabolomic analyses will further enable the investigation of diet-gene interactions, supporting the development of precision nutrition strategies for individuals at elevated genetic risk. This research is expected to inform strategies for disease prevention and the maintenance of functional independence in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 years or older.
* Volunteers of the Tzu Chi Foundation.
* Participating in the 2-day comprehensive health examination program.

Exclusion Criteria:

* Pregnant individual.
* Diagnosed with dementia or poor cognition resulting in inability to answer questionnaires.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Middle-aged and older adults (≥40 years) who are volunteers of the Tzu Chi Foundation or their relatives and friends, participating in the 2-day comprehensive health examination program in Taiwan.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive Function | From enrollment to three-year follow-up, six-year follow up
  Cognitive function will be assessed using Montreal Cognitive Assessment [MoCA], Taiwanese version. (Score range 0-30, unit = points). A score ≥26 is generally considered normal, while scores <26 suggest possible cognitive impairment. Outcomes will be reported both as continuous MoCA scores and as a binary classification (normal vs. impaired).
Appendicular skeletal muscle mass | From baseline to three-year follow-up, six-year follow-up
  Appendicular skeletal muscle mass (ASM) will be assessed by bioimpedance analysis (BIA), with height-adjusted cutoffs of <7.0 kg/m² in men and <5.7 kg/m² in women defined as low ASM. Results will be reported as both continuous measures (kg/m²) and categorical measures (normal or low ASM).
Grip strength | From baseline to three-year follow-up, six-year follow-up
  Grip strength will be assessed using a handheld dynamometer, with cutoffs defined as <28 kg for men and <18 kg for women. Results will be reported as continuous measures (kg).
Sarcopenia | From baseline to three-year follow-up, six-year follow-up
  Sarcopenia will be defined as the combined presence of low ASM and low grip strength. Results will be reported as a binary outcome (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Hsueh-Ting Chiu, PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (1):
- Dalin Tzu Chi Hospital., Dalin, Chiayi, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided